CLINICAL TRIAL: NCT00508313
Title: Phase I Assessment of Thermal Signature of Patients Undergoing Radiation Therapy
Brief Title: Thermal Signature of Patients Undergoing Radiation Therapy
Status: Withdrawn | Type: Observational
Why Stopped: Study closed early without enrollment.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-1082
Record Dates: First submitted 2007-07-26; First posted 2007-07-27 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2009-09

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Healthy Control; Thermal Imaging; Thermal Signatures; Radiation Therapy; Chemoradiation Therapy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With Lung Cancer: Patients with lung cancer.
  Interventions: Procedure: Thermal Imaging
- Healthy Participants: Healthy participants without cancer.
  Interventions: Procedure: Thermal Imaging

INTERVENTIONS:
Procedure: Thermal Imaging — Thermal imaging sessions, each taking approximately 10 minutes.

SUMMARY:
The goal of this clinical research study is to evaluate whether thermal imaging (recording body temperature) can be used to check the body's response to cancer therapy.

Primary Objective:

* The primary objective of this study is to establish techniques and methodologies of quantifying thermal signatures and their changes for cancer patients undergoing chemoradiation therapy.

Secondary Objective:

* The secondary objective is to evaluate correspondence between changes of thermal signature of a normal organ, e.g. lung or esophagus, versus the toxicity of that organ from chemoradiation therapy.

DETAILED DESCRIPTION:
For Patients:

THERMAL IMAGER:

A thermal imager (a camera similar to a digital camera) takes pictures of skin surfaces. The imager is able to view temperature distribution of the skin surface.

STUDY PARTICIPATION:

If you agree to take part in this study, your body temperature will be measured with thermal imaging.

You will have thermal imaging sessions several times before the cancer treatment starts and during the therapy course. You will be given detailed instructions on how to prepare for the imaging sessions ahead of time as well as what to expect during the imaging sessions.

Before beginning thermal imaging, your temperature will be measured with a thermometer. To perform thermal imaging, you will be asked to take off all of your clothes in a private room and stand still in front of a thermal imaging camera. No one will be present while you disrobe. When you have finished taking off your clothes a radiation oncologist or other medical doctor will record several pictures from a computer stationed outside the room. Pictures of your front, back, and side views will be taken. These pictures will look like a silhouette (body outline) with thermal coloring. The entire imaging session should take about 10 minutes to complete each time.

LENGTH OF STUDY:

Your participation will be over in this study after the thermal images have been recorded.

This is an investigational study. Thermal imaging is FDA approved and commercially available for breast cancer screening. Its use in this study is investigational. Up to 35 patients will take part in this study. All will be enrolled at M. D. Anderson.

For Volunteers:

THERMAL IMAGER:

A thermal imager (a camera similar to a digital camera) takes pictures of skin surfaces. The imager is able to view temperature distribution of the skin surface.

STUDY PARTICIPATION:

If you agree to take part in this study, your body temperature will be measured with thermal imaging.

You will have thermal imaging sessions several times during the course of this study. You will be given detailed instructions on how to prepare for the imaging sessions ahead of time as well as what to expect during the imaging sessions.

Before beginning thermal imaging, your temperature will be measured with a thermometer. To perform thermal imaging, you will be asked to take off all of your clothes in a private room and stand still in front of a thermal imaging camera. No one will be present while you disrobe. When you have finished taking off your clothes a radiation oncologist or other medical doctor will record several pictures from a computer stationed outside the room. Pictures of your front, back, and side views will be taken. These pictures will look like a silhouette (body outline) with thermal coloring. The entire imaging session should take about 10 minutes to complete each time.

Volunteers will not participate in any part of cancer treatment, diagnostic imaging tests (CT, PET, etc), or any other clinical procedures in MD Anderson. Volunteers will not need to see physicians at MD Anderson or elsewhere. Thermal images will be taken 4 times during one day for a volunteer (morning, midmorning, earlier afternoon, late afternoon). Volunteers should not take any medications or perform any other medical procedures from morning to late afternoon until the thermal imaging is completed.

LENGTH OF STUDY:

Your participation will be over in this study after the thermal images have been recorded.

This is an investigational study. Thermal imaging is FDA approved and commercially available for breast cancer screening. Its use in this study is investigational. Up to 10 volunteers without cancer (5 males and 5 non-pregnant females) will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with lung cancers of any stages.
2. Patients will undergo chemotherapy or radiation therapy.
3. Patients with KPS > 70, are physically mobile and independent, and are able to stand still straight for more than 10 minutes for imaging purposes.
4. Age >18 years

Exclusion Criteria:

1. Patients who had lung surgery within past 3 months.
2. Patients with breast implant or cardiac implant (pace maker or defibrillator).
3. Patients who had skin diseases (e.g. skin desquamation, dermatitis) or other medical conditions that may interfere with thermal measurement.
4. Pregnant woman
5. Extreme obese patients with body mass index >=35

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer and healthy participants without cancer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Change in Participant Thermal Signature as determined by Thermal imaging (recording body temperature) | Imaging session takes about 10 minutes to complete each time, imaging beginning at baseline and continuing till 12 months post therapy, up to 24 months
  Body temperature at the time of the thermal imaging taken using a commercial infrared camera; thermal imaging sessions several times before the cancer treatment starts, during and after the radiotherapy courses. Using thermal images taken from multiple sessions, both the absolute and relative changes of the temperature distribution will be calculated and analyzed. The location of the regions will be guided by the diagnostic computed tomography (CT) and Positron Emission Positron emission tomography (PET)/CT images for temperatures at multiple angles of body, site of radiation for skin reaction, primary cancer site and critical normal organs.

SECONDARY OUTCOMES:
Number Toxicities Experienced by Participants according to CTCAE v. 3.0 | Baseline to 24 months
  Chemoradiation related toxicity, including hematological and nonhematological acute and late side effects assessed during each clinic visit and follow up session including patient clinical symptoms and clinical assessment of treatment-related toxicity as assessed by NCI Common Terminology Criteria for Adverse Events version 3.0 (CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: Zhongxing Liao, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org